CLINICAL TRIAL: NCT03452228
Title: A Phase 2, Randomized, Placebo-Controlled Study of Safety and Efficacy, Following Repeat-Dose Administration of Evinacumab (Anti-ANGPTL3) in Patients With Severe Hypertriglyceridemia (sHTG) at Risk for Acute Pancreatitis
Brief Title: Safety and Efficacy Following Repeat-Dose of Evinacumab (Anti-ANGPTL3) in Patients With Severe Hypertriglyceridemia (sHTG) at Risk for Acute Pancreatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1500-HTG-1522; 2016-003307-62 (EudraCT Number)
Record Dates: First submitted 2018-01-30; First posted 2018-03-02 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Severe Hypertriglyceridemia (sHTG)
MeSH Terms: conditions — Hypertriglyceridemia | interventions — evinacumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- evinacumab (Experimental)
  Interventions: Drug: evinacumab
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: evinacumab — Administered by Intravenous (IV)
  Other Names: REGN1500
  Arms: evinacumab
Drug: Placebo — Administered by Intravenous (IV)
  Arms: Placebo

SUMMARY:
The primary objective is to determine the change in Triglyceride (TG) levels following 12 weeks of repeated Intravenous (IV) doses of evinacumab.

ELIGIBILITY:
Key Inclusion Criteria:

1. Previous documentation in the patient's medical records of a fasting serum TG measurement ≥ 1000 mg/dL (11.3 mmol/L) on more than 1 occasion, and all fasting TG values ≥500 mg/dL (5.6 mmol/L) at screening
2. History of a hospitalization and diagnosis of acute pancreatitis in the past 10 years
3. On stable lipid-modifying diet with or without medications (eg, statins, niacin, omega-3 fatty acids). Lipid-modifying diet and doses of medications should be stable for at least 4 weeks (6 weeks for fibrates, 8 weeks for PCSK9 inhibitors) prior to screening
4. Body mass index (BMI) of 18-40 kg/m2

Key Exclusion Criteria:

1. A hospital or clinic discharge diagnosis of acute pancreatitis within 12 weeks of screening
2. Lipid apheresis or plasma exchange treatment within the last 4 weeks or plans to undergo apheresis or plasma exchange during the time frame of the study
3. History of class 3/4 heart failure at any time in the past, or hospitalization for heart failure, diagnosis of a myocardial infarction, stroke, Transient ischemic attack (TIA), unstable angina, Coronary artery bypass surgery (CABG), Percutaneous coronary intervention (PCI), carotid surgery/stenting within 3 months before the screening visit
4. History of bleeding disorders, esophageal varices, heparin induced thrombocytopenia, or contraindications to receiving heparin (eg, allergic reaction to heparin)
5. Previous treatment with Glybera® in the past 5 years or treatment with lomitapide or mipomersen in the past 6 months
6. Pregnant or breast feeding women

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (16):
- United States (9):
  - Regeneron Research Facility, Boca Raton, Florida
  - Regeneron Research Facility, Atlanta, Georgia
  - Regeneron Research Facility, Kansas City, Kansas
  - Regeneron Research Facility, New York, New York
  - Regeneron Research Facility, Philadelphia, Pennsylvania
  - Regeneron Research Facility, Pittsburgh, Pennsylvania
  - Regeneron Research Facility, Dallas, Texas
  - Regeneron Research Facility, Houston, Texas
  - Regeneron Research Facility, Milwaukee, Wisconsin
- Canada (2):
  - Regeneron Research Facility, Chicoutimi, Quebec
  - Regeneron Research Facility, Québec, Quebec
- Italy (2):
  - Regeneron Research Facility, Napoli, Campania
  - Regeneron Research Facility, Rome
- United Kingdom (3):
  - Regeneron Research Facility, Birmingham
  - Regeneron Research Facility, London
  - Regeneron Research Facility, Manchester

REFERENCES:
- [Derived] Rosenson RS, Gaudet D, Ballantyne CM, Baum SJ, Bergeron J, Kershaw EE, Moriarty PM, Rubba P, Whitcomb DC, Banerjee P, Gewitz A, Gonzaga-Jauregui C, McGinniss J, Ponda MP, Pordy R, Zhao J, Rader DJ. Evinacumab in severe hypertriglyceridemia with or without lipoprotein lipase pathway mutations: a phase 2 randomized trial. Nat Med. 2023 Mar;29(3):729-737. doi: 10.1038/s41591-023-02222-w. Epub 2023 Mar 6. PMID 36879129

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 centers enrolled participants in Italy, Canada, the United Kingdom of Great Britain and Northern Ireland, and the United States.
Pre-assignment Details: Based upon information (or lack of information) on genotype in medical history at screening, eligible patients were enrolled into 1 of 3 cohorts; 51 of 74 patients screened were randomized and treated during the double-blind treatment period (DBTP).
Groups:
- Placebo IV Q4W (DBTP): Participants received placebo matching evinacumab intravenously (IV) every 4 weeks (Q4W) on days 1, 29, and 57 during 12-week DBTP.
- Evinacumab 15 mg/kg (DBTP): Participants received IV infusion of evinacumab 15 milligram per kilogram (mg/kg) Q4W on days 1, 29, and 57 during the 12-week DBTP.
- Evinacumab 15 mg/kg (SBTP): All participants who completed the DBTP (placebo IV Q4W and evinacumab 15 mg/kg arm) received IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141 during 12-week the SBTP.
Period: Double-Blind Treatment Period (12 Weeks)
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg (DBTP) | Evinacumab 15 mg/kg (SBTP)
Started (Randomized) | 17 | 35 | 0
Treated (Randomized and Treated) | 16 | 35 | 0
Actual Cohort 1 (Actual Cohort 1 included participants with homozygous or compound heterozygous loss-of-function (LOF) mutations in genes in the lipoprotein lipase (LPL) pathway as was determined based on genotype data.) | 5 | 12 | 0
Actual Cohort 2 (Actual Cohort 2 included participants with heterozygous LOF mutations in genes in the LPL pathway as was determined based on genotype data.) | 6 | 9 | 0
Actual Cohort 3 (Actual Cohort 3 included participants without LOF mutations in genes in the LPL pathway as was determined based on genotype data.) | 5 | 14 | 0
Completed | 15 | 32 | 0
Not Completed | 2 | 3 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Randomized but not treated | 1 | 0 | 0
Period: Single-Blind Treatment Period (12 Weeks)
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg (DBTP) | Evinacumab 15 mg/kg (SBTP)
Started | 0 | 0 | 47 (Participants were moved from DBTP to SBTP.)
Treated | 0 | 0 | 47
Actual Cohort 1: DB Placebo to SB Evinacumab (Actual Cohort 1 included participants with homozygous or compound heterozygous LOF mutations in genes in the LPL pathway as was determined based on genotype data. Those actual cohort 1 participants who received placebo in DBTP were shifted into single blind (SB) evinacumab group.) | 0 | 0 | 4
Actual Cohort 1: DB Evinacumab to SB Evinacumab (Actual Cohort 1 included participants with homozygous or compound heterozygous LOF mutations in genes in the LPL pathway as was determined based on genotype data. Those actual cohort 1 participants who received evinacumab in DBTP were shifted into SB evinacumab group.) | 0 | 0 | 11
Actual Cohort 2: DB Placebo to SB Evinacumab (Actual Cohort 2 included participants with heterozygous LOF mutations in genes in the LPL pathway as was determined based on genotype data. Those actual cohort 2 participants who received placebo in DBTP were shifted into SB evinacumab group.) | 0 | 0 | 6
Actual Cohort 2: DB Evinacumab to SB Evinacumab (Actual Cohort 2 included participants with heterozygous LOF mutations in genes in the LPL pathway as was determined based on genotype data. Those actual cohort 2 participants who received evinacumab in DBTP were shifted into SB evinacumab group.) | 0 | 0 | 9
Actual Cohort 3: DB Placebo to SB Evinacumab (Actual Cohort 3 included participants without LOF mutations in genes in the LPL pathway as was determined based on genotype data. Those actual cohort 3 participants who received placebo in DBTP were shifted into SB evinacumab group.) | 0 | 0 | 5
Actual Cohort 3: DB Evinacumab to SB Evinacumab (Actual Cohort 3 included participants without LOF mutations in genes in the LPL pathway as was determined based on genotype data. Those actual cohort 3 participants who received evinacumab in DBTP were shifted into SB evinacumab group.) | 0 | 0 | 12
Completed | 0 | 0 | 43
Not Completed | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received any double-blind study drug based on the treatment assigned (as randomized).
Groups:
- Placebo IV Q4W (DBTP): Participants received placebo matching evinacumab IV Q4W on days 1, 29, and 57 during 12-week DBTP.
- Evinacumab 15 mg/kg (DBTP): Participants received IV infusion of evinacumab 15 mg/kg Q4W on days 1, 29, and 57 during the 12-week DBTP.
- Total: Total of all reporting groups
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg (DBTP) | Total
Number analyzed (Participants) | 16 | 35 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (13.10) | 48.6 (10.23) | 47.8 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 17 | 24
  Male | 9 | 18 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 14 | 31 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 5 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 12 | 29 | 41
    Other | 3 | 0 | 3
Fasting Triglycerides [Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)] | 2303.8 (1503.81) | 2475.1 (1597.20) | 2421.4 (1555.50)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG) Level Following 12 Weeks of Repeated IV Doses of Evinacumab in Actual Cohort 3 Participants
Description: For participants randomized to evinacumab treatment group, baseline (Week 0) TG was defined as the geometric mean of all available TG results at day -28, day -14 and week 0; for participants randomized to placebo treatment group, baseline (Week 12) TG was defined as the geometric mean of all available TG results at weeks 6, 8, and 12.
Time Frame: Participants randomized to evinacumab: Week 0 corresponds to Baseline and 12 weeks treatment corresponds to Week 12 of the DBTP; Participants randomized to placebo: Week 12 corresponds to Baseline and 12 weeks treatment corresponds to Week 24 of the SBTP
Population: The FAS included all randomized participants who received any double-blind study drug based on the treatment assigned (as randomized). Mixed-effect Model for Repeated Measures (MMRM) method assessed within-patient treatment comparisons (using an unstructured covariance matrix), while accounting for baseline TG, study visit, and baseline TG by study visit interaction. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Groups:
- Actual Cohort 3: DB Placebo/SB Evinacumab IV 15mg/kg Q4W: Participants without LOF mutations in genes in the LPL pathway as was determined based on genotype data received placebo matched to evinacumab on days 1, 29, and 57 in 12-week DBTP and were shifted to 12-week SBTP, to receive IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141.
- Actual Cohort 3: DB Evinacumab/SB Evinacumab IV 15mg/kg Q4W: Participants without LOF mutations in genes in the LPL pathway as was determined based on genotype data received evinacumab 15 mg/kg Q4W on days 1, 29, and 57 in 12-week DBTP and were shifted to 12-week SBTP, to receive IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141.
Arm/Group | Actual Cohort 3: DB Placebo/SB Evinacumab IV 15mg/kg Q4W | Actual Cohort 3: DB Evinacumab/SB Evinacumab IV 15mg/kg Q4W
Number analyzed (Participants) | 5 | 14
Percent Change | 19.2 (99.1) | -37.2 (42.9)
Statistical Analysis 1: Comparison: Actual Cohort 3: DB Placebo/SB Evinacumab IV 15mg/kg Q4W; Test type: Superiority; Median Difference (Final Values) = -43.5, 95% CI 2-sided [-89.4 to 1238.9]
Statistical Analysis 2: Comparison: Actual Cohort 3: DB Evinacumab/SB Evinacumab IV 15mg/kg Q4W; Test type: Superiority; Median Difference (Final Values) = -75.5, 95% CI 2-sided [-82.2 to 121.2]

2. Secondary Outcome: Percent Change From Baseline in Fasting TG Level Following 2 to 24 Weeks of Repeated IV Doses of Evinacumab Overall Group
Description: Percent change from baseline in fasting TG level following 2 to 24 weeks of repeated IV doses of evinacumab overall group during DBTP and SBTP was reported.
Time Frame: DBTP: Baseline, Weeks 2, 4, 6, 8, 12; SBTP: Weeks 16, 20, and 24
Population: The FAS included all randomized participants who received any double-blind study drug based on the treatment assigned (as randomized). Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure for specified arm/period and "number analyzed" signifies to participants evaluable for this outcome at given timepoints.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Placebo Q4W (DBTP): Participants received placebo matching evinacumab IV Q4W on days 1, 29, and 57 during the 12-week DBTP.
- Evinacumab IV 15mg/kg Q4W (DBTP): Participants received IV infusion of evinacumab 15 mg/kg Q4W on days 1, 29, and 57 during the 12-week DBTP.
- Evinacumab IV 15mg/kg Q4W (SBTP): All participants who completed the DBTP (placebo IV Q4W and evinacumab 15 mg/kg arms) received IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141 during 12-week SBTP.
Arm/Group | Placebo Q4W (DBTP) | Evinacumab IV 15mg/kg Q4W (DBTP) | Evinacumab IV 15mg/kg Q4W (SBTP)
Number analyzed (Participants) | 16 | 32 | 47
Percent Change
  Percent change at Week 2: number analyzed (Participants) | 16 | 31 | 0
  Percent change at Week 2 | 1.99 (45.687) | -51.38 (33.160) |
  Percent change at Week 4: number analyzed (Participants) | 14 | 32 | 0
  Percent change at Week 4 | -3.52 (41.029) | -43.70 (39.119) |
  Percent change at Week 6: number analyzed (Participants) | 15 | 31 | 0
  Percent change at Week 6 | 92.56 (262.368) | -52.69 (40.214) |
  Percent change at Week 8: number analyzed (Participants) | 14 | 32 | 0
  Percent change at Week 8 | 4.83 (38.941) | -32.86 (64.787) |
  Percent change at Week 12: number analyzed (Participants) | 14 | 32 | 0
  Percent change at Week 12 | 17.47 (47.610) | -42.03 (61.086) |
  Percent change at Week 16: number analyzed (Participants) | 0 | 0 | 46
  Percent change at Week 16 |  |  | -39.23 (46.026)
  Percent change at Week 20: number analyzed (Participants) | 0 | 0 | 46
  Percent change at Week 20 |  |  | -38.09 (49.070)
  Percent change at Week 24: number analyzed (Participants) | 0 | 0 | 47
  Percent change at Week 24 |  |  | -35.86 (65.011)

3. Secondary Outcome: Percent Change From Baseline in Fasting TG Level Following 2 to 24 Weeks of Repeated IV Doses of Evinacumab in Actual Cohorts 1, 2, and 3
Description: Percent change from baseline in fasting TG level following 2 to 24 weeks of repeated IV doses of evinacumab in actual cohorts 1, 2, and 3 participants were reported.
Time Frame: Weeks 2, 4, 6, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent Change
Groups:
- Actual Cohort 1: DB Evinacumab/SB Evinacumab IV 15mg/kg Q4W: Participants with homozygous or compound heterozygous LOF mutations in genes in the LPL pathway as was determined based on genotype data received evinacumab 15 mg/kg Q4W on days 1, 29, and 57 in 12-week DBTP and were shifted to 12-week SBTP, to receive IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141.
- Actual Cohort 2: DB Evinacumab/SB Evinacumab IV 15mg/kg Q4W: Participants with heterozygous LOF mutations in genes in the LPL pathway as was determined based on genotype data received evinacumab 15 mg/kg Q4W on days 1, 29, and 57 in 12-week DBTP and were shifted to 12-week SBTP, to receive IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141.
Arm/Group | Actual Cohort 1: DB Evinacumab/SB Evinacumab IV 15mg/kg Q4W | Actual Cohort 2: DB Evinacumab/SB Evinacumab IV 15mg/kg Q4W | Actual Cohort 3: DB Evinacumab/SB Evinacumab IV 15mg/kg Q4W
Number analyzed (Participants) | 12 | 9 | 14
Percent Change
  Percent change at Week 2: number analyzed (Participants) | 11 | 9 | 11
  Percent change at Week 2 | -28.3 [-40.3 to -6.5] | -77.5 [-81.2 to -58.9] | -74.4 [-84.2 to -37.1]
  Percent change at Week 4: number analyzed (Participants) | 11 | 9 | 12
  Percent change at Week 4 | -19.0 [-69.6 to -2.7] | -48.0 [-76.2 to -29.2] | -70.3 [-83.4 to -50.2]
  Percent change at Week 6: number analyzed (Participants) | 11 | 9 | 11
  Percent change at Week 6 | -47.1 [-59.1 to -5.6] | -84.6 [-85.7 to -61.3] | -71.3 [-87.0 to -39.5]
  Percent change at Week 8: number analyzed (Participants) | 11 | 9 | 12
  Percent change at Week 8 | -29.5 [-72.0 to 4.8] | -69.2 [-72.2 to -58.4] | -62.5 [-84.8 to 48.0]
  Percent change at Week 12: number analyzed (Participants) | 11 | 9 | 12
  Percent change at Week 12 | -27.7 [-68.5 to 2.2] | -64.8 [-84.5 to -41.8] | -81.7 [-90.5 to -21.7]
  Percent change at Week 16: number analyzed (Participants) | 11 | 9 | 12
  Percent change at Week 16 | -16.2 [-56.7 to 29.3] | -71.3 [-80.8 to -57.1] | -80.4 [-87.2 to -37.3]
  Percent change at Week 20: number analyzed (Participants) | 11 | 9 | 12
  Percent change at Week 20 | -37.2 [-49.9 to -8.8] | -65.5 [-70.2 to -45.8] | -75.7 [-88.1 to -6.6]
  Percent change at Week 24: number analyzed (Participants) | 11 | 9 | 12
  Percent change at Week 24 | -7.7 [-31.8 to 9.1] | -75.7 [-82.3 to -57.1] | -71.4 [-86.5 to -54.0]

4. Secondary Outcome: Change From Baseline in Total Score of Participants Reported Abdominal and Gastrointestinal (GI) Symptoms Using Hypertriglyceridemia and Acute Pancreatitis Symptom Scale (HAP-SS)
Description: HAP-SS: 19-item measure of symptoms with a 24-hour recall period. 4 pain items were captured on 0-10-point severity NRS, each scored 0 (No pain) to 10 (Worst possible pain), while 15 non-pain items captured on 5-point frequency Likert scale, each scored from 1 (None of the time) to 5 (All of the time). Pain domain 4 items: stomach pain average, worst stomach pain, worst back pain, stomach pain after eating (score range: 0 to 40). Abdominal symptoms domain 6 items: bloated, nausea, vomiting, passed excessive gas, diarrhea, light-colored or greasy stool (score range: 6 to 30). Physical symptoms domain 5 items: fever, insomnia, excessive sweating, dizziness, racing heart rate (score range 5 to 25). Other symptoms domain 4 items: fatigue, loss of appetite, hungry after eating, felt full after eating a small amount (score range 4 to 20). All items were transformed on to total score ranges from 0 (no symptoms) to 100 (severe symptoms). Negative change indicates better condition.
Time Frame: Baseline, Week 12 (DBTP), Week 24 (SBTP)
Population: Patient-reported outcomes (PRO) analysis set included all randomized participants who received any double-blind study treatment with a baseline and at least 1 non-missing post-baseline PRO evaluation. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure for specified arm/period.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Placebo IV Q4W (DBTP): Participants received placebo matching evinacumab IV Q4W on days 1, 29, and 57 during the 12-week DBTP.
- Evinacumab IV 15mg/kg (DBTP): Participants received IV infusion of evinacumab 15 mg/kg Q4W on days 1, 29, and 57 during the 12-week DBTP.
- Evinacumab IV 15mg/kg (SBTP): All participants who completed the DBTP (placebo IV Q4W and evinacumab 15 mg/kg arms) received IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141 during 12-week SBTP.
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab IV 15mg/kg (DBTP) | Evinacumab IV 15mg/kg (SBTP)
Number analyzed (Participants) | 12 | 23 | 28
Score on a Scale
  DBTP: Change at Week 12: number analyzed (Participants) | 12 | 23 | 0
  DBTP: Change at Week 12 | -0.69 (6.930) | -0.74 (5.102) |
  SBTP: Change at Week 24: number analyzed (Participants) | 0 | 0 | 28
  SBTP: Change at Week 24 |  |  | -0.12 (5.033)

5. Secondary Outcome: Change From Baseline in Total Score of Participants Reported Dietary Behavior Questionnaire (HAP-DB)
Description: Dietary habits and impact were measured by the Hypertriglyceridemia and Acute Pancreatitis Dietary Behavior (HAP-DB) questionnaire, a 6- item measure of dietary behavior that had a 24-hour recall period using a 5-point frequency Likert scale (1= None of the time to 5= All of the time) and a dietary impact total score, ranging from 6 (no impact) to 30 (severe impact). The six HAP-DB items were: 1 -amount of food eaten), 2 -fatty or greasy food), 3 -carbohydrates), i4 (-sugar or sugary foods), 5 -alcohol intake), 6 -skipped meal). The total score was calculated as the sum of the six item scores and then transformed to a 0-100 score, where lower score indicates less of an issue with dietary behaviors. Transformed score = 100 * (score - minimum possible score) / (maximum - minimum possible score). Change from baseline in total score of participants reported daily dietary habits and impact questionnaire during DBTP and SBTP was reported.
Time Frame: Baseline, Week 12 (DBTP), Week 24 (SBTP)
Population: PRO analysis set includes all randomized participants who received any double-blind study treatment with a baseline and at least 1 non-missing post-baseline PRO evaluation. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure for specified arm/period.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab IV 15mg/kg (DBTP) | Evinacumab IV 15mg/kg (SBTP)
Number analyzed (Participants) | 12 | 23 | 28
Score on a Scale
  DBTP: Change at Week 12: number analyzed (Participants) | 12 | 23 | 0
  DBTP: Change at Week 12 | -2.267 (5.5897) | 2.021 (15.2152) |
  SBTP: Change at Week 24: number analyzed (Participants) | 0 | 0 | 28
  SBTP: Change at Week 24 |  |  | -1.255 (7.7864)

6. Secondary Outcome: DBTP: Change From Baseline in Degree of Pancreatic Injury/Inflammation Through 18F-2-Fluoro-2-Deoxy-D Glucose Positron Emission Tomography (18F-FDG-PET) Imaging Following 12 Weeks of Treatment With Evinacumab Assessed by 18F-FDG SUVmax and SUVmean
Description: 18F-FDG-PET is a molecular imaging modality that has demonstrated high sensitivity in the in vivo detection of glycolytic tissues, including tumors and inflammatory foci. 18F-FDG PET has been applied in a clinical setting to the assessment of inflammation for a variety of indications, including auto immune pancreatitis, atherosclerosis and infection. 18F-FDG-PET was performed at baseline (placebo run-in period) and following 12 weeks of study treatment (double-blind treatment period) as a method to measure inflammation in the pancreas. Here, SUVmax was standardized uptake values maximum and SUVmean was mean standardized uptake values were reported.
Time Frame: as for outcome 1
Population: PET analysis set included all randomized participants who received any double-blind study treatment with a baseline and a post-baseline (positron emission tomography) PET evaluation. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure for specified arm/period.
Measure: Mean (Standard Deviation); unit: gram/milliliter (g/ml)
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab IV 15mg/kg Q4W (DBTP)
Number analyzed (Participants) | 12 | 25
gram/milliliter (g/ml)
  SUVmax: Baseline | 2.318 (0.6168) | 2.738 (0.6027)
  SUVmax: Change at Week 12 | 0.576 (1.0628) | 0.185 (0.5830)
  SUVmean: Baseline | 1.212 (0.2513) | 1.478 (0.2000)
  SUVmean: Change at Week 12 | 0.175 (0.2117) | -0.007 (0.2312)

7. Secondary Outcome: DBTP: Change From Baseline in Degree of Pancreatic Injury/Inflammation Through Diffusion Weighted-Magnetic Resonance Imaging (DW-MRI) Following 12 Weeks of Treatment With Evinacumab Assessed by Apparent Diffusion Coefficient (ADC)
Description: In DW-MRI the random diffusion of water molecules occurring within intracellular, extracellular and intravascular spaces were measured, enabling detection of macroscopic soft tissue pathology such as edema, necrosis and fibrosis. The ADC was a principal metric quantified in DW-MRI experiments, where ADC values was mapped across a region of interest at a spatial resolution of ~3*3*5 cubic millimeter (mm^3). Normal pancreas ADCs were considered as (1.77±0.32)*103 square-millimeters per second (mm^2/sec) while acute pancreatitis ADCs were (1.32±0.32)* 103 mm^2/sec showing a significant window for measuring projected inflammatory changes in pancreas. DW-MRI was performed at baseline (placebo run-in period) and following 12 weeks of study treatment (double-blind treatment period) as a method to measure inflammation in the pancreas. Change from baseline in degree of pancreatic injury/inflammation through DW-MRI following 12 weeks of treatment with evinacumab assessed by ADC was reported.
Time Frame: as for outcome 1
Population: Magnetic resonance imaging (MRI) analysis set included all randomized participants who received any double-blind study treatment with a baseline and at least 1 post-baseline MRI evaluation. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure for specified arm/period and "number analyzed" signifies to participants evaluable for this outcome at given timepoints.
Measure: Mean (Standard Deviation); unit: Square-millimeters per second (mm^2/sec)
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab IV 15mg/kg Q4W (DBTP)
Number analyzed (Participants) | 14 | 28
Square-millimeters per second (mm^2/sec)
  DBTP: Baseline | 0.00144 (0.000303) | 0.00154 (0.000257)
  DBTP: Change at Week 12: number analyzed (Participants) | 13 | 26
  DBTP: Change at Week 12 | -0.00007 (0.000107) | 0.00001 (0.000133)

8. Secondary Outcome: SBTP: Change From Baseline to Degree of Pancreatic Injury/Inflammation Through DW-MRI Following 24 Weeks of Treatment With Evinacumab as Assessed by ADC
Description: In DW-MRI, the random diffusion of water molecules occurring within intracellular, extracellular and intravascular spaces were measured, enabling detection of macroscopic soft tissue pathology such as edema, necrosis and fibrosis. The ADC was a principal metric quantified in DW-MRI experiments, where ADC values was mapped across a region of interest at a spatial resolution of ~3*3*5 mm^3. Normal pancreas ADCs were considered as (1.77±0.32)*103 mm^2/sec while acute pancreatitis ADCs are (1.32±0.32)* 103 mm^2/sec showing a significant window for measuring the projected inflammatory changes in the pancreas. Change from baseline to degree of pancreatic injury/inflammation through DW-MRI following 24 weeks of treatment with evinacumab assessed by ADC was reported.
Time Frame: Baseline (Week 0 DBTP), Week 24 (SBTP)
Population: MRI analysis set included all randomized participants who received any double-blind study treatment with a baseline and at least 1 post-baseline MRI evaluation. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure for specified arm/period.
Measure: Mean (Standard Deviation); unit: mm^2/sec
Arm/Group | Evinacumab IV 15mg/kg Q4W (SBTP)
Number analyzed (Participants) | 37
mm^2/sec | -0.00001 (0.000166)

9. Secondary Outcome: Total Evinacumab Concentration in Serum
Description: Concentrations of total evinacumab in serum by time and DBTP treatment group reported
Time Frame: Up to 44 weeks
Population: Pharmacokinetic (PK) analysis set included all randomized participants who received any study drug and have at least 1 non-missing measurement of evinacumab concentration following the first dose of the study drug. Here, "number analyzed" signifies to participants evaluable for this outcome at given timepoints.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Groups:
- Placebo IV Q4W (DBTP): Participants received placebo matching evinacumab IV Q4W on days 1, 29, and 57 during the 12-week DBTP. Participants were then shifted to 12-week SBTP, to receive IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141.
- Evinacumab IV 15mg/kg Q4W (DBTP): Participants received IV infusion of evinacumab 15 mg/kg Q4W on days 1, 29, and 57 during the 12-week DBTP. Participants were then shifted to 12-week SBTP, to receive IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141.
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab IV 15mg/kg Q4W (DBTP)
Number analyzed (Participants) | 16 | 35
milligram per liter (mg/L)
  Week 0: Pre-Dose | NA (NA) — Value below the limit of quantification | NA (NA) — Value below the limit of quantification
  Week 0: End Of Infusion: number analyzed (Participants) | 16 | 34
  Week 0: End Of Infusion | 24.3 (97.0) | 561 (203)
  Week 4: Pre-Dose: number analyzed (Participants) | 14 | 31
  Week 4: Pre-Dose | NA (NA) — Value below the limit of quantification | 73.6 (38.3)
  Week 4: End of Infusion: number analyzed (Participants) | 14 | 30
  Week 4: End of Infusion | 0.334 (1.25) | 590 (153)
  Week 8: Pre-Dose: number analyzed (Participants) | 13 | 31
  Week 8: Pre-Dose | NA (NA) — Value below the limit of quantification | 109 (57.2)
  Week 8: End of Infusion: number analyzed (Participants) | 13 | 32
  Week 8: End of Infusion | 28.8 (104) | 586 (119)
  Week 12: Pre-Dose: number analyzed (Participants) | 14 | 31
  Week 12: Pre-Dose | 0.00639 (0.0239) | 124 (81.4)
  Week 12: End Of Infusion: number analyzed (Participants) | 13 | 32
  Week 12: End Of Infusion | 544 (159) | 662 (146)
  Week 20: Pre-Dose: number analyzed (Participants) | 14 | 32
  Week 20: Pre-Dose | 113 (51.9) | 160 (119)
  Week 20: End Of Infusion: number analyzed (Participants) | 14 | 32
  Week 20: End Of Infusion | 675 (146) | 680 (199)
  Week 24: Post Last Dose 4 Weeks: number analyzed (Participants) | 15 | 32
  Week 24: Post Last Dose 4 Weeks | 121 (76.7) | 134 (77.2)
  Week 28: Post Last Dose 8 Weeks: number analyzed (Participants) | 12 | 28
  Week 28: Post Last Dose 8 Weeks | 43.1 (47.8) | 40.2 (44.6)
  Week 36: Post Last Dose 16 Weeks: number analyzed (Participants) | 10 | 23
  Week 36: Post Last Dose 16 Weeks | 0.239 (0.250) | 1.98 (7.41)
  Week 44: Post Last Dose 24 Weeks: number analyzed (Participants) | 12 | 27
  Week 44: Post Last Dose 24 Weeks | 0.0190 (0.0464) | 0.0680 (0.102)

10. Secondary Outcome: Total Angiopoietin-like (ANGPTL3) Concentration in Serum
Description: Concentrations of total ANGPTL3 in serum by time and DBTP treatment group reported
Time Frame: Up to 44 weeks
Population: The total target analysis set is defined as all randomized participants who received any study drug and have at least 1 non-missing measurement of total ANGPTL3 concentration following the first dose of study drug. Here, "number analyzed" signifies to participants evaluable for this outcome at given timepoints.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab IV 15mg/kg Q4W (DBTP)
Number analyzed (Participants) | 16 | 35
mg/L
  Week 0: Pre-Dose | 0.0929 (0.0313) | 0.105 (0.0327)
  Week 0: End of Infusion: number analyzed (Participants) | 16 | 34
  Week 0: End of Infusion | 0.0950 (0.0256) | 0.258 (0.0745)
  Week 4: Pre-Dose: number analyzed (Participants) | 14 | 31
  Week 4: Pre-Dose | 0.111 (0.0272) | 0.265 (0.0932)
  Week 4: End of Infusion: number analyzed (Participants) | 14 | 30
  Week 4: End of Infusion | 0.106 (0.0205) | 0.404 (0.132)
  Week 8: Pre-Dose: number analyzed (Participants) | 13 | 31
  Week 8: Pre-Dose | 0.114 (0.0333) | 0.307 (0.0758)
  Week 8: End of Infusion: number analyzed (Participants) | 13 | 32
  Week 8: End of Infusion | 0.137 (0.0977) | 0.415 (0.0875)
  Week 12: Pre-Dose: number analyzed (Participants) | 14 | 31
  Week 12: Pre-Dose | 0.107 (0.0273) | 0.310 (0.0911)
  Week 12: End of Infusion: number analyzed (Participants) | 13 | 32
  Week 12: End of Infusion | 0.250 (0.0940) | 0.394 (0.102)
  Week 20: Pre-Dose: number analyzed (Participants) | 14 | 32
  Week 20: Pre-Dose | 0.302 (0.0973) | 0.346 (0.101)
  Week 20: End of Infusion: number analyzed (Participants) | 14 | 32
  Week 20: End of Infusion | 0.407 (0.144) | 0.422 (0.118)
  Week 24: Post Last Dose 4 Weeks: number analyzed (Participants) | 15 | 32
  Week 24: Post Last Dose 4 Weeks | 0.294 (0.0954) | 0.331 (0.113)
  Week 28: Post Last Dose 8 Weeks: number analyzed (Participants) | 12 | 28
  Week 28: Post Last Dose 8 Weeks | 0.311 (0.0701) | 0.265 (0.0984)
  Week 36: Post Last Dose 16 Weeks: number analyzed (Participants) | 10 | 23
  Week 36: Post Last Dose 16 Weeks | 0.134 (0.0487) | 0.193 (0.0969)
  Week 44: Post Last Dose 24 Weeks: number analyzed (Participants) | 12 | 27
  Week 44: Post Last Dose 24 Weeks | 0.107 (0.0322) | 0.131 (0.0489)

11. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADA)
Description: ADA were classified as the following: 1) Negative any time (negative in ADA assay at all time points); 2) Pre-existing immunoreactivity (ADA positive response at baseline with all post treatment ADA results negative or ADA positive response at baseline with all post treatment responses less than 9-fold of baseline titer levels); 3) Treatment-boosted Response (ADA positive response in assay post first dose that is at least 9-fold over baseline titer levels, when baseline results were positive); 4) Treatment-emergent ADA response (ADA positive response post first dose, when baseline results were negative or missing). Number of participants with ADA by DBTP treatment group reported.
Time Frame: Up to 44 weeks
Population: The ADA analysis set included all randomized participants who received any study drug and had at least 1 non-missing ADA result following the first dose of study treatment. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure for specified arm/period.
Measure: Count of Participants; unit: Participants
Groups:
- Evinacumab 15 mg/kg IV (DBTP): Participants received IV infusion of evinacumab 15 mg/kg Q4W on days 1, 29, and 57 during the 12-week DBTP. Participants were then shifted to 12-week SBTP, to receive IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141.
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg IV (DBTP)
Number analyzed (Participants) | 15 | 34
Participants
  Negative any Time | 14 | 29
  Pre-existing Immunoreactivity | 1 | 4
  Treatment-boosted Response | 0 | 0
  Treatment-emergent Response | 0 | 1

12. Secondary Outcome: DBTP: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: TEAEs are AEs that developed or worsened or became serious during the respective TEAE period. Number of participants who experienced a TEAE/serious TEAE during the DBTP reported.
Time Frame: From first dose of DB treatment to day of last dose of DB treatment + 24 weeks (if not proceeding to SBTP) or up to day before first dose of SB treatment in SBTP
Population: The double-blind safety analysis set considered for safety analyses included the randomized population who received at least 1 dose or part of a dose of double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg (DBTP)
Number analyzed (Participants) | 16 | 35
Participants
  Participants with at least one TEAE | 11 | 25
  Participants with at least one serious TEAE | 3 | 4

13. Secondary Outcome: SBTP: Number of Participants With TEAEs and Serious TEAEs
Description: TEAEs are AEs that developed or worsened or became serious during the respective TEAE period. Number of participants who experienced a TEAE/serious TEAE during the SBTP reported.
Time Frame: From day of first SB study treatment to day of last SB treatment + 24 weeks
Population: The single-blind safety analysis set considered for safety analyses included the randomized population who received at least 1 dose or part of a dose of single-blind study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Evinacumab 15 mg/kg (SBTP): All participants who completed the DBTP (placebo IV Q4W and evinacumab 15 mg/kg arms) received IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141 during 12-week SBTP.
Arm/Group | Evinacumab 15 mg/kg (SBTP)
Number analyzed (Participants) | 47
Participants
  Participants with at least one TEAE | 38
  Participants with at least one Serious TEAE | 15

14. Secondary Outcome: Number of Participants With Liver Function Laboratory Abnormalities in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP), and Total Bilirubin
Description: The number of participants with laboratory abnormalities in ALT, AST, ALP, and total bilirubin that fell into the pre-defined potentially clinically significant value (PCSV) categories reported: ALT: greater than (>)2 upper limit of normal (ULN) and baseline (BL) less than or equal to (<=) 2 ULN, less than (>) 3 ULN and baseline <= 3 ULN, >5 ULN and baseline <= 5 ULN, >10 ULN and baseline ≤ 10 ULN, >20 ULN and baseline <= 20 ULN; AST: >2 ULN and baseline ≤ 2 ULN, >3 ULN and baseline <= 3 ULN, >5 ULN and baseline <= 5 ULN, >10 ULN and baseline <= 10 ULN, >20 ULN and baseline <= 20 ULN; ALP: > 1.5 ULN and baseline <= 1.5 ULN; Total Bilirubin (TB): > 1.5 ULN and baseline <= 1.5 ULN, > 2 ULN and baseline <= 2 ULN.
Time Frame: Baseline up to 44 weeks
Population: The double-blind safety analysis set considered for safety analyses included the randomized population who received at least 1 dose or part of a dose of double-blind study drug. The single-blind safety analysis set considered for safety analyses included the randomized population who received at least 1 dose or part of a dose of single-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg (DBTP) | Evinacumab 15 mg/kg (SBTP)
Number analyzed (Participants) | 16 | 35 | 47
Participants
  ALT >2 ULN and <=3 ULN and <=2 ULN at baseline: number analyzed (Participants) | 16 | 34 | 47
  ALT >2 ULN and <=3 ULN and <=2 ULN at baseline | 0 | 1 | 0
  ALT >3 ULN and <=5 ULN and <=3 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  ALT >3 ULN and <=5 ULN and <=3 ULN at BL | 0 | 2 | 0
  ALT >5 ULN and <=10 ULN and <=5 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  ALT >5 ULN and <=10 ULN and <=5 ULN at BL | 0 | 0 | 2
  ALT 10 ULN and <=20 ULN and <=10 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  ALT 10 ULN and <=20 ULN and <=10 ULN at BL | 0 | 0 | 0
  ALT >20 ULN and <=20 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  ALT >20 ULN and <=20 ULN at BL | 0 | 0 | 0
  AST >2 ULN and <=3 ULN and <=2 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  AST >2 ULN and <=3 ULN and <=2 ULN at BL | 0 | 2 | 0
  AST >3 ULN and <=5 ULN and <=3 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  AST >3 ULN and <=5 ULN and <=3 ULN at BL | 0 | 1 | 1
  AST >5 ULN and <=10 ULN and <=5 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  AST >5 ULN and <=10 ULN and <=5 ULN at BL | 0 | 0 | 1
  AST >10 ULN and <=20 ULN and <=10 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  AST >10 ULN and <=20 ULN and <=10 ULN at BL | 0 | 0 | 0
  AST >20 ULN and <=20 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  AST >20 ULN and <=20 ULN at BL | 0 | 0 | 0
  Bilirubin >1.5 ULN - <=2 ULN and =<1.5 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  Bilirubin >1.5 ULN - <=2 ULN and =<1.5 ULN at BL | 0 | 0 | 0
  Bilirubin >2 ULN and =< 2.0 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  Bilirubin >2 ULN and =< 2.0 ULN at BL | 0 | 0 | 0
  Alkaline Phosphatase >1.5 ULN and =< 1.5 ULN at BL: number analyzed (Participants) | 16 | 34 | 47
  Alkaline Phosphatase >1.5 ULN and =< 1.5 ULN at BL | 0 | 0 | 2
  (ALT>3ULN&TB>2ULN)&(ALT<=3ULN or TB<=2ULN) at BL: number analyzed (Participants) | 16 | 33 | 47
  (ALT>3ULN&TB>2ULN)&(ALT<=3ULN or TB<=2ULN) at BL | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to Last Single-Blind (SB) dose + 168 days (24 weeks), up to approximately 44 weeks
Groups:
- Placebo IV Q4W (DBTP): Participants received placebo matching evinacumab IV Q4W) on days 1, 29, and 57 during the 12-week DBTP.
- Evinacumab 15 mg/kg (SBTP): All participants who completed the DBTP received IV infusion of evinacumab 15 mg/kg Q4W on days 85, 113, and 141 during 12-week in the SBTP.
- SBTP DB/SB Evinacumab IV 15mg/kg Q4W: Participants received evinacumab 15 mg/kg IV Q4W on days 1, 29, and 57 during the 12-week DBTP. During the 12-week SBTP, participants continued to receive evinacumab 15 mg/kg IV Q4W on days 85, 113, and 141.
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg (DBTP) | Evinacumab 15 mg/kg (SBTP) | SBTP DB/SB Evinacumab IV 15mg/kg Q4W
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/35 | 0/15 | 0/32
Serious Adverse Events (participants affected / at risk) | 3/16 | 4/35 | 4/15 | 11/32
Other Adverse Events (participants affected / at risk) | 11/16 | 20/35 | 13/15 | 22/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV Q4W (DBTP) (N=16) | Evinacumab 15 mg/kg (DBTP) (N=35) | Evinacumab 15 mg/kg (SBTP) (N=15) | SBTP DB/SB Evinacumab IV 15mg/kg Q4W (N=32)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4) | 8 (14)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV Q4W (DBTP) (N=16) | Evinacumab 15 mg/kg (DBTP) (N=35) | Evinacumab 15 mg/kg (SBTP) (N=15) | SBTP DB/SB Evinacumab IV 15mg/kg Q4W (N=32)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (6) | 2 (3) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03452228/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03452228/SAP_001.pdf